CLINICAL TRIAL: NCT04715893
Title: Ostomy Belt Use Associated Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Vanessa Hui, Assistant Professor of Clinical Surgery, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20201333
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-02

CONDITIONS: Stoma Ileostomy; Stoma Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ostomy belt group (Experimental): Participants in this group will receive ostomy belts for eight weeks.
  Interventions: Other: Ostomy belt

INTERVENTIONS:
Other: Ostomy belt — Stealth ostomy belt continuous for eight weeks

SUMMARY:
The objective of this study is to elucidate whether the use of an ostomy belt can improve the quality of life in patients with an ostomy.

ELIGIBILITY:
Inclusion Criteria:

* Current patients at University of Miami Hospital with stoma willing to trial an ostomy belt
* 18 - 70 years old
* Willing and able to sign informed consent

Exclusion Criteria:

* Patients without stoma or unwilling to wear ostomy belt.
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Change in quality of life as measured by SQOLS | Baseline to 4 weeks, baseline to 8 weeks post ostomy belt use
  Quality of life will be assessed using the Stoma Quality of Life Scale questionnaire (SQOLS) with a range in score from 0 to 100 in overall satisfaction in life with a higher score indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Hui, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No